CLINICAL TRIAL: NCT04741984
Title: The DEMAND Study: Dose Escalation Study of Monocyte Antigen Carrier Cells for Newly Diagnosed Glioblastoma With Unmethylated MGMT Gene Promoter
Brief Title: Monocyte Antigen Carrier Cells for Newly Diagnosed GBM
Acronym: DEMAND
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to need to proceed with procedural changes with goals of improving the technical and economic feasibility.
Sponsor: Michael Gunn (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Michael Gunn, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105363; 5P01CA225622 (NIH)
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Glioblastoma; Glioma, Malignant
Keywords: DEMAND; Desjardins; Pro00105363; Glioblastoma; Vaccine; Duke; Gunn; 20211706
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MT-201-GBM monocyte vaccine (Experimental): pp65 monocyte vaccines (MT-201-GBM) - cohorts of patients will receive increasing doses (dose escalation) of MT-201-GBM followed by a dose expansion cohort at the maximum tolerated dose. Patients will receive a total of 3 intravenous vaccines every 4 weeks after completing standard radiation therapy (XRT) and temozolomide (TMZ) and a single course of dose-intensified TMZ.
  Interventions: Biological: MT-201-GBM monocyte vaccine

INTERVENTIONS:
Biological: MT-201-GBM monocyte vaccine — monocytes isolated from patient's leukapheresis loaded with CMV pp65-LAMP (Lysosomal-associated Membrane Protein) mRNA (Messenger Ribonucleic Acid)

SUMMARY:
The primary purpose of this study is to determine the maximum tolerated dose (MTD) of MT-201-GBM (pp65CMV antigen monocytes) that will be administered to patients newly diagnosed with a type of brain tumor called glioblastoma (GBM) that has an unmethylated MGMT (O[6]-methylguanine-DNA methyltransferase) (MGMT) gene promoter.

DETAILED DESCRIPTION:
The investigational vaccine (MT-201-GBM) in this study is made from a type of immune cell called monocytes, which have been engineered to express a cytomegalovirus (CMV) protein.

The monocyte vaccines are made from the patient's own cells, which are collected through a procedure called leukapheresis. During leukapheresis, the patient's blood is collected into a machine that removes white blood cells and then returns the remainder of the blood back to the individual. The leukapheresis procedure is not typically associated with any discomfort or pain. The white blood cells collected from leukapheresis are used to generate the patient's monocyte vaccine. After leukapheresis, patients receive standard radiation therapy combined with temozolomide for about 6 weeks, followed by one cycle of temozolomide for 21 days. About 2 days later, patients will receive the first monocyte vaccine, followed by 2 more monocyte vaccines every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age;
* Newly diagnosed glioblastoma patient with definitive resection prior to enrollment, with residual radiographic contrast enhancement on most recent magnetic resonance imaging (MRI) of <1 cm in maximal diameter in any axial plane;
* Able to receive SOC XRT/TMZ for approximately 6 weeks duration and of more than 54GY;
* MRI post XRT does not show progressive disease outside the radiation field;
* Karnofsky Performance Status (KPS) score ≥ 70%;
* MGMT promoter unmethylated (Determined by Caris Life Science pyrosequencing);
* Hemoglobin ≥ 9.0 g/dl, absolute neutrophil count (ANC) ≥ 1,000 cells/µl, platelets ≥ 100,000 cells/µl prior to starting TMZ cycle 1 (patient must meet these criteria within 4 weeks after the end of XRT/TMZ to be eligible);
* Serum creatinine ≤ 3 times institutional upper limit of normal (ULN) for age, serum aspartate aminotransferase (AST) ≤ 3 times institutional ULN for age;
* Bilirubin ≤ 1.5 times ULN prior to starting TMZ cycle 1 (Exception: Patient has known Gilbert's Syndrome or patient has suspected Gilbert's Syndrome, for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.)
* Signed informed consent approved by the Institutional Review Board (IRB);
* Female patients must not be pregnant or breast-feeding. Female patients of childbearing potential (defined as < 2 years after last menstruation or not surgically sterile) must use a highly effective contraceptive method (allowed methods of birth control, [i.e. with a failure rate of < 1% per year] are implants, injectables, combined oral contraceptives, intra-uterine device [IUD], sexual abstinence or vasectomized partner) during the trial and for a period of at least 6 months following the last administration of trial drug(s). Female patients with an intact uterus (unless amenorrhea for the last 24 months) must have a negative serum pregnancy test within 48 hours prior to first study treatment.
* Fertile male patients must agree to use a highly effective contraceptive method (allowed methods of birth control [i.e. with a failure rate of < 1% per year] include a female partner using implants, injectables, combined oral contraceptives, IUDs, sexual abstinence or prior vasectomy) during the trial and for a period of at least 6 months following the last administration of trial drugs.

Exclusion Criteria:

* Pregnant or breast-feeding;
* Women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception;
* Patients with known potentially anaphylactic allergic reactions to gadolinium-DTPA (diethylenetriamine penta-acetic acid);
* Patients who cannot undergo MRI;
* Patients with evidence of tumor in the brainstem, cerebellum, or spinal cord, radiological evidence of multifocal disease, or leptomeningeal disease;
* Patients who cannot tolerate TMZ;
* Severe, active comorbidity, including any of the following:

  * Unstable angina and/or congestive heart failure requiring hospitalization;
  * Transmural myocardial infarction within the last 6 months;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of study initiation;
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy;
  * Known hepatic insufficiency resulting in clinical jaundice and/or coagulation defects;
  * Known HIV positive status, Hepatitis B, Hepatitis C;
  * Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy;
  * Active connective tissue disorders, such as lupus or scleroderma that, in the opinion of the treating physician, may put the patient at high risk for radiation toxicity;
* Co-medication that may interfere with study results (e.g., immuno-suppressive agents other than corticosteroids);
* Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin (Treatment with tamoxifen or aromatase inhibitors or other hormonal therapy that may be indicated in prevention of prior cancer disease recurrence are not considered current active treatment.)
* Current, recent (within 4 weeks of the administration of this study agent), or planned participation in an experimental drug study;
* Patients are not permitted to have had any other conventional therapeutic intervention other than steroids prior to enrollment outside of standard of care chemotherapy and radiation therapy. Patients who receive previous inguinal lymph node dissection, radiosurgery, brachytherapy, or radiolabeled monoclonal antibodies will be excluded.
* Known history of autoimmune disease (with the exceptions of medically-controlled hypothyroidism and Type I Diabetes Mellitus);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of MT-201-GBM | 1 month after first infusion
  Dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate of 0.25.
pp65 T-cell Immune Response After 2 Weeks Post Infusion Three Compared to Baseline | 2 weeks after third infusion
  Mean (or median) change from baseline within each dose level for IFN gamma, granzyme-B, and fluorospot

SECONDARY OUTCOMES:
Percentage of patients with a dose-limiting toxicity (DLT) during DLT observation period within each dose level | 1 month after first infusion
  To assess safety and tolerability of MT-201-GMB, the percentage of patients with a dose-limiting toxicity (DLT) during the DLT observation period within each dose level will be estimated.
Median Overall Survival (OS) | 2 years
  Survival from start of MT-201-GBM
Median Progression Free Survival (PFS) | 2 years
  Time to first recurrence after start of MT-201-GBM
pp65 T-cell Immune Response After Each Infusion Compared to Baseline | 2 weeks after third infusion
  Mean (or median) change from baseline to peak levels within each dose level for IFN gamma and ELISpot

CONTACTS AND LOCATIONS:
Overall Officials: Annick S Desjardins, MD, FRCPC, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — http://tischbraintumorcenter.duke.edu/
- See also: Duke Health — http://www.dukehealth.org/clinical-trials